CLINICAL TRIAL: NCT02263664
Title: Observational Study of Sublingual Microcirculatory Blood Flow Characteristics in Patients Undergoing Transthoracic Esophagectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Randal Blank, MD, Associate Professor, Anesthesiology, University of Virginia
Other Study IDs: 17551
Record Dates: First submitted 2014-09-08; First posted 2014-10-13 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Transthoracic Esophagectomy
Keywords: microcirculation; esophagectomy; side stream dark field; microcirculatory derangements

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Microcirculatory alterations occur in critically ill patients and those undergoing major surgeries. The severity of perioperative microvascular alterations appear to be related to the severity of organ dysfunction after surgery. Non-cardiac thoracic surgeries comprise a subgroup of high risk surgical procedures which have the potential to significantly affect and impair microcirculatory function but this patient population has not been well studied. Esophagectomy surgery in particular produces a profound systemic inflammatory response which correlates with a number of adverse outcomes. It is likely, though unproven, that microcirculatory derangements may underly these phenomena. Though the study of microcirculatory dysfunction in thoracic surgery is in its infancy, the body of available evidence at this point supports the following hypotheses; that microcirculatory derangements and dysfunction 1) occur during major surgeries including transthoracic esophagectomy 2) may be related to SIRS, 3) may predict adverse outcomes, and 4) may be amenable to modification via specific therapies.

We propose a prospective observational study to determine the effects of transthoracic esophagectomy on microcirculatory function. Two hundred patients meeting inclusion criteria undergoing planned transthoracic esophagectomy via thoracotomy incision will be prospectively enrolled at The University of Virginia. Patients will be followed for 28 days or until discharge from the ICU. Evaluation of the sublingual, gastric serosal and mucosal tissues will be performed using sidestream dark field (SDF) imaging using the CytoCam® by Braedius Medical BV (Huizen, The Netherlands). Scoring of the microcirculation will include an index of vascular density (perfused vessel density), an assessment of capillary perfusion (proportion of perfused vessels and microcirculatory flow index) and a heterogeneity index.

Note: the CytoCam® will only take a series of images as consistent with a microscope of exposed tissue. Also, the FDA Office of Device Evaluations (ODE) General Surgery Devices Branch One - Light Based/laser (GSDB1) has deemed this device to be exempt from 510(K) approval.

http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfPCD/classification.cfm?ID=5021

Data from patient's medical charts before and after surgery (30 days post) will be used for elucidation of specific complications. We will use the cardiovascular and respiratory components of the SOFA score as independent measures of organ dysfunction. Acute kidney injury will be defined by the AKIN criteria as an increase of at least 50% above baseline serum creatinine and will be graded from stage 1 to 3.

DETAILED DESCRIPTION:
1. Provide the scientific background, rationale and relevance of this project. The microcirculation plays a fundamental role in gas and nutrient exchange; it must constantly adapt by controlling vascular tone and regional blood flow. In disease states, increased permeability may be necessary to produce the inflammatory response. The assessment and quantification of the macrovascular hemodynamics and the assumption that it is reflective of microvascular change is fundamentally flawed. Even when global hemodynamic variables are corrected, many patients with circulatory failure will develop multi organ failure and ultimately die. The recent advent of in vivo microcirculation monitoring has begun to improve our understanding of the relationships between surgery, anesthetic management, and regulation of the microcirculation.

Microcirculatory alteration also occurs in patients undergoing cardiac surgery. Bauer et al first reported that microcirculatory perfusion was transiently altered in humans after cardiopulmonary bypass. Similar findings were reported more recently by other groups. , More importantly, these alterations can also be observed in patients who undergo surgery without cardiopulmonary bypass.3 Furthermore the sublingual microcirculation was still slightly abnormal up to 24 h after surgery in these patients. As in non-cardiac surgery, the severity of perioperative microvascular alterations correlated with peak lactate levels and severity of organ dysfunction after surgery.iii High-risk surgery is a new area in which in vivo microcirculatory alterations have been observed. In patients undergoing high-risk non-cardiac surgery, Jhanji et al observed that the density and proportion of perfused capillaries was lower in the 14 patients who subsequently developed postoperative complications than in the 11 patients with an uneventful postoperative course. Subcutaneous tissue PO2 and laser Doppler cutaneous blood flow did not differ between the groups, further highlighting the lack of sensitivity of these methods to detect heterogeneous perfusion. Interestingly, there was no significant difference in global O2 delivery between the groups.

Non-cardiac thoracic surgeries comprise a subgroup of high risk surgical procedures which have the potential to significantly affect and impair microcirculatory function. A study of patients undergoing esophagectomy demonstrated significant impairment of sublingual microcirculation relative to pancreaticoduodenectomy patients. Esophagectomy surgery produces a profound systemic inflammatory response which correlates to a number of adverse outcomes. Interestingly, the time course of microcirculatory impairment and recovery appears to parallel the SIRS typically seen in surgeries of this type. Transthoracic esophagectomy is typically facilitated by one lung ventilation (OLV) in an effort to optimize surgical exposure to the operative hemithorax. The institution of OLV has the potential to dramatically impair tissue oxygen supply demand relationships via adverse effects on systemic oxygen desaturation, as a result of an increased venous admixture from right to left intrapulmonary shunting, as well as decrements in cardiac output. Cerebral oxygen desaturation accompanying OLV is also well described, though the pathophysiology is not well understood. It is likely, though unproven, that microcirculatory derangements may underly these phenomena. Though the study of microcirculatory dysfunction in thoracic surgery is in its infancy, the body of available evidence at this point supports the following hypotheses; that microcirculatory derangements and dysfunction 1) occur during major surgeries including transthoracic esophagectomy 2) may be related to SIRS, OLV or both, 3) may predict adverse outcomes, and 4) may be amenable to modification via specific therapies.

This is a feasibility study to see if the changes in microcirculatory parameters as observed by the SDF device can accurately diagnose anastomotic and other complications for the purpose of leading to a wider study of microcirculatory derangements as an indicator of risk of surgical complications.

Hypothesis to be Tested:

i. Microcirculatory derangements, as indicated by changes in microcirculation of sublingual tissue, serosa tunica near the surgical division, or the mucosal lining of the stomach near the surgical division, occur during transthoracic esophagectomy and in the perioperative period.

ii. Changes in microcirculation predicts post-operative anastomotic complications iii. Changes in microcirculation predicts post-operative complications

Specific Aims

1. Determine whether microcirculatory derangements, as indicated by changes in microcirculation of sublingual tissue, serosa tunica near the surgical division, or the mucosal lining of the stomach near the surgical division, occur during transthoracic esophagectomy involving one lung ventilation (OLV), using a side stream dark field (SDF) imaging system.

   1.1. This aim will include measurements of microcirculatory parameters at multiple time points within the perioperative period.
2. Determine the temporal relationship of microcirculatory dysfunction and recovery, if any, at the initiation of OLV, reestablishment of two lung ventilation, and cessation of surgery.

   2.1. This aim will include measurements of microcirculatory parameters at multiple time points within the perioperative period.
3. Determine whether observed changes in microcirculation is predictive of postoperative organ dysfunction, and perioperative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 through 75 years
2. Subjects are undergoing transthoracic esophagectomy utilizing thoracotomy or thoracoscopy incisions as part of their clinical care. These surgeries include primarily the Ivor Lewis, and three hole (McKeown) esophagectomy procedures and variants thereof.
3. A patent arterial line
4. A patent IV line
5. Must be able to read and speak English
6. Subjects may have current diagnosis of cancer that requires esophagectomy as part of their clinical care.

Exclusion Criteria:

1. Subjects unable/unwilling to give informed consent.
2. Cognitively Impaired
3. Prisoners
4. Pregnant females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Race: ANY
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Microcirculation parameters as observed with Sidestream Dark Field Microscopy an indicator of post operative complications | 3 YEARS
  Is Microcirculation derangement in the mucosal bed an indicator of post-operative complications? Can we use the Sidestream Dark Field Microscopy to detect microcirculation derangements as a precursor to post operative complications?

CONTACTS AND LOCATIONS:
Overall Officials: RANDAL BLANK, M.D. PH.D, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Bauer A, Kofler S, Thiel M, Eifert S, Christ F. Monitoring of the sublingual microcirculation in cardiac surgery using orthogonal polarization spectral imaging: preliminary results. Anesthesiology. 2007 Dec;107(6):939-45. doi: 10.1097/01.anes.0000291442.69337.c9. PMID 18043062
- [Background] Atasever B, Boer C, Goedhart P, Biervliet J, Seyffert J, Speekenbrink R, Schwarte L, de Mol B, Ince C. Distinct alterations in sublingual microcirculatory blood flow and hemoglobin oxygenation in on-pump and off-pump coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2011 Oct;25(5):784-90. doi: 10.1053/j.jvca.2010.09.002. Epub 2010 Nov 5. PMID 21115363
- [Background] Koning NJ, Vonk AB, Meesters MI, Oomens T, Verkaik M, Jansen EK, Baufreton C, Boer C. Microcirculatory perfusion is preserved during off-pump but not on-pump cardiac surgery. J Cardiothorac Vasc Anesth. 2014 Apr;28(2):336-41. doi: 10.1053/j.jvca.2013.05.026. Epub 2013 Oct 23. PMID 24161555
- [Background] Jhanji S, Lee C, Watson D, Hinds C, Pearse RM. Microvascular flow and tissue oxygenation after major abdominal surgery: association with post-operative complications. Intensive Care Med. 2009 Apr;35(4):671-7. doi: 10.1007/s00134-008-1325-z. Epub 2008 Oct 21. PMID 18936911
- [Background] van Genderen M, Gommers D, Klijn E, Lima A, Bakker J, van Bommel J. Postoperative sublingual microcirculatory derangement following esophagectomy is prevented with dobutamine. Clin Hemorheol Microcirc. 2011;48(4):275-83. doi: 10.3233/CH-2011-1421. PMID 22012833
- [Background] Wright CD, Kucharczuk JC, O'Brien SM, Grab JD, Allen MS; Society of Thoracic Surgeons General Thoracic Surgery Database. Predictors of major morbidity and mortality after esophagectomy for esophageal cancer: a Society of Thoracic Surgeons General Thoracic Surgery Database risk adjustment model. J Thorac Cardiovasc Surg. 2009 Mar;137(3):587-95; discussion 596. doi: 10.1016/j.jtcvs.2008.11.042. PMID 19258071